CLINICAL TRIAL: NCT02851446
Title: Prevalence and Risk Factors of Dreentilation Syndrome in a Population of Patients Under Ventilation for Whatever Reason
Brief Title: Prevalence and Risk Factors of Reventilation Syndrome in a Population of Patients Under Ventilation for Whatever Reason
Acronym: DEVENTILATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: FOIGNOT 2015
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Prevalence of and Factors Associated With Reventilation Syndrome (DS)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- DS
  Interventions: Other: measure dyspnoea> Borg 7
- no DS
  Interventions: Other: measure dyspnoea> Borg 7

INTERVENTIONS:
Other: measure dyspnoea> Borg 7

SUMMARY:
Non-invasive nocturnal ventilation is an effective treatment for chronic respiratory failure, whether due to obstructive (COPD), restrictive or neuromuscular causes, notably for patients in the last two categories for whom it significantly prolongs life expectancy. Overall, the treatment is well tolerated, its principal adverse effects being discomfort related to the mask.

In certain patients, morning dyspnoea when the mask is removed has been described. This is disabling as it limits everyday activities for at least 30 minutes, and defines deventilation syndrome. The pathophysiology of this syndrome is uncertain, notably the roles of hyperinflation, patient/ventilator asynchrony, or the sudden increase in diaphragmatic work after a night of rest.

The aim of this study is to investigate the prevalence of and factors associated with reventilation syndrome (DS) in a population of patients with ventilation whatever the reason, in a stable state, and followed by the medical devices department of Dijon CHU, so as to better understand the mechanisms. Patients with DS will subsequently be invited to participate in a therapeutic trial.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* ventilation for whatever reason
* in the ST mode
* not in life support
* at more than 1 month after the last episode of respiratory decompensation

Exclusion Criteria:

* guardianship
* inability to understand instructions and provide consent
* uncontrolled psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population of patients with ventilation whatever the reason, in a stable state, and followed by the medical devices department of Dijon CHU
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
presence of diagnostic criteria for reventilation Syndrome (dyspnoea > Borg 7) | at withdrawal of the machine, disabling for everyday activities for at least 30 minutes after stopping the ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France